CLINICAL TRIAL: NCT01196156
Title: An Observational Phase IV Study for Prospective Follow-up to Adult Height of a Cohort of Subjects Born Small for the Gestational Age and Treated With Growth Hormone
Brief Title: Follow-up to Adult Height of a Cohort of Subjects Born Small for the Gestational Age and Treated With Growth Hormone
Acronym: SGA
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck, S.L., Spain (Industry)
Responsible Party: Sponsor
Other Study IDs: IMP 27143
Record Dates: First submitted 2010-08-26; First posted 2010-09-08 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Infant, Small for Gestational Age
Keywords: Infant, Small for Gestational Age; Dwarfism Pituitary; Saizen; Somatropin; Growth Hormone; Insulin resistance
MeSH Terms: conditions — Dwarfism, Pituitary; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This non-interventional study for prospective follow up of a cohort of 220 subjects born small for gestational age (SGA) is planned for the purpose of finding out if normalisation of adult height is associated or not with metabolic alterations and if true, their magnitude and relevance as well as to detect warnings throughout the treatment period that may be useful for prevention or therapy. This study would help in answering the question if the SGA and growth hormone (GH) association results in insulin resistance and if affirmative, who develops it as well as its impact on other metabolic parameters that precedes type 2 diabetes.

DETAILED DESCRIPTION:
The small for gestational age (SGA) concept includes babies born to term whose weight and/or height is lower than two standard deviations (SD) below the mean. Pathologically short stature is understood as a stature of 2.5 SD below the mean for their age and an expected adult height adjusted to the parental height of one SD below the mean. These SGA children with a pathological short stature after four years of age are unsuitable for GH treatment. In fact, there is no other efficient treatment for short stature and insufficient development of these children other than GH. In addition to short stature, the SGA syndrome also includes resistance to insulin with the consequent risk of developing type 2 diabetes and other interrelated metabolic alterations like dyslipidemia and hypertension; and the glucose-insulin-insulin growth factors (IGFs)-proteins transport axis regulate growth as well as foetal metabolism and development. Independent from the possible maternal environmental causes, those born with SGA have low levels of somatomedin C (IGF-I) and its transport protein [Insulin-like growth factor binding protein 3 (IGFBP-3)] as well as fasting hyperinsulinemia. The low levels of IGF-1 and IGFBP-3 persist in those that do not present a catch-up growth and the insulin resistance is secondary to the somatotrope axis. Treatment with GH increases IGF-I and IGFBP3 levels but also the plasmatic level of fasting insulin and the long term net result of this combination is unknown.

An analysis has shown, that although during the first 2 years of GH treatment, there are no signs of glucose intolerance even though there is less sensitivity to insulin, there could be a greater incidence of type 2 diabetes in deficient children that have been treated with GH for a longer period. Treatment with GH, of children born SGA that have not caught-up their growth at 4 years of age, in the majority of cases achieves a good initial growth speed increase in order to continue to grow within normal limits and end up with an adult height that falls within normal. This is achieved with an authorised daily dose of 0.035 mg/kg (1 mg/m2/day). However, the question regarding the possible metabolic consequences of GH treatment of those born SGA remains unanswered in both forms, to find out if GH treatment increases or reduces resistance to insulin and other associated metabolic parameters and therefore, the risk of developing type 2 diabetes. Continued monitoring to adult height of a cohort of subjects born with SGA and treated with GH is the most efficient, easy and comfortable tool for answering that question.

OBJECTIVES

Primary objective:

* To quantify the evolution of insulin sensitivity from the start of treatment with GH until adult stature is reached. Sensitivity or resistance to insulin is calculated using the HOMA-IR model (Homeostasis Model Assessment for Insulin Resistance) which is a reliable and easy mathematical model that uses the following formula: insulinemia (μU/ml) x glycemia (mmol/l)/22.5.

Secondary objectives:

* To find predictive factors for the possible changes in insulin sensitivity and its complex associated obesity, hypertension and high triglycerides type dyslipidemia with low high density lipoprotein (HDL)-cholesterol. For this, a relation between these metabolic factors and auxological parameters is to be identified.

  a. The following are considered independent or predictive variables:
* Speed of growth in cm/ year
* Standard deviations of height
* IGF-I in ng/ml
* IGFBP-3 in ng/ml b. The dependent variables will be:
* HOMA-IR value
* Triglycerides rate in mg/dl / HDL-cholesterol in mg/dl
* Blood pressure in mmHG
* Body mass index

This is an observational study of a single cohort, without the possibility of a control group because those born with SGA, who experience a catch-up growth and enter normal auxology within the first four years of life are not subjected to a paediatric follow-up similar to those that do not catch-up to normal auxology and are treated with GH. Therefore, the same auxological and metabolic test results are not available in standard care. The collection of said parameters requires an "ad hoc" intervention and the study would be experimental or interventional. The observation period of this study encompasses from the start of treatment with GH up to a year after finishing the treatment for any reason. The starting age as well as the time treatment is ended will vary per subject. However, most subjects finish treatment once adulthood is reached. In accordance with clinical studies, the average observation period will probably be about 10 years. After the basal data is made available, the collection of data afterwards will be carried out once a year per subject.

ELIGIBILITY:
Inclusion Criteria:

* Children with growth disorder (current height <-2.5 SD and height adjusted to parental stature <-1 SD) in children born SGA with a weight and/or length at birth below -2 SD, that has not experimented a growth catch-up (growth speed <0 SD during the last year) at 4 years old or afterwards were enrolled in the study
* Children undergoing treatment with somatropin from Serono
* Children whose parent or legal guardians, as well as the subject himself if 12 or more years old have given written permission to access their records

Exclusion Criteria:

* Children with closed epiphysis
* Children with known hypersensitivity to somatropin or to any excipients present in the injection powder or solvent
* Subjects with active neoplasms. Any anti-tumoral treatment must be completed prior to starting treatment with somatropin
* Subjects with evidence of progression or relapse of a subjacent intracranial lesion
* Subjects with acute critical diseases such as those that present complications after open heart surgery, abdominal surgery, polytraumatisms, acute respiratory failure or similar conditions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children with growth disorder (current height <-2.5 SD and height adjusted to parental stature <-1 SD) in children born SGA with a weight and/or length at birth below -2 SD, that has not experimented a growth catch-up (growth speed <0 SD during the last year) at 4 years old or afterwards.
Sampling Method: Non-Probability Sample
Enrollment: 443 (Actual)
Dates: Start 2005-09-30 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in the insulin sensitivity index measured using HOMA-IR (Homeostasis Model Assessment for Insulin Resistance) | up to 10 years
  Once a year per subject from the start of treatment with GH up to a year after finishing the treatment for any reason

SECONDARY OUTCOMES:
Auxological parameter - Growth speed | up to 10 years
  Growth speed will be measured using a wall stadiometer and quantified and assessed in cm/year. Measurement occurs once a year per subject from the start of treatment with GH up to a year after finishing the treatment for any reason.
Auxological parameter - Height | up to 10 years
  Height will be measured using a wall stadiometer and quantified in standard deviations (SDS). Measurement occurs once a year per subject from the start of treatment with GH up to a year after finishing the treatment for any reason.
Auxological parameter - Weight in kilogram | up to 10 years
  Measurement occurs once a year per subject from the start of treatment with GH up to a year after finishing the treatment for any reason.
Auxological parameter - Plasma insulin growth factor (IGF-I), measured at the local laboratory | up to 10 years
  Plasma IGF-1 will be quantified in ng/ml. Measurement occurs once a year per subject from the start of treatment with GH up to a year after finishing the treatment for any reason.
Auxological parameter - Plasma insulin growth factor (IGF-I), measured at the central laboratory | up to 10 years
  Plasma IGF-1 will be quantified in ng/ml. Measurement occurs once a year per subject from the start of treatment with GH up to a year after finishing the treatment for any reason.
Metabolic parameter - Fasting plasma insulin measured at the local laboratory | up to 10 years
  Fasting plasma insulin will be quantified in μU/ml. Measurement occurs once a year per subject from the start of treatment with GH up to a year after finishing the treatment for any reason.
Metabolic parameter - Fasting plasma glucose measured at the local laboratory | up to 10 years
  Fasting plasma insulin will be quantified in mmol/l. Measurement occurs once a year per subject from the start of treatment with GH up to a year after finishing the treatment for any reason.
Metabolic parameter - Plasma triglycerides measured locally | up to 10 years
  Plasma triglycerides will be quantified in mg/dl. Measurement occurs once a year per subject from the start of treatment with GH up to a year after finishing the treatment for any reason.
Metabolic parameter - High density lipoproteins (HDL) cholesterol measured locally | up to 10 years
  HDL-cholesterol will be quantified in mg/dl. Measurement occurs once a year per subject from the start of treatment with GH up to a year after finishing the treatment for any reason.
Metabolic parameter - Glycosylated haemoglobin (HbA1c) | up to 10 years
  HbA1c will be quantified in % over total Hb. Measurement occurs once a year per subject from the start of treatment with GH up to a year after finishing the treatment for any reason.
Metabolic parameter - Blood pressure (BP) | up to 10 years
  BP will be measured in mmHg. Measurement occurs once a year per subject from the start of treatment with GH up to a year after finishing the treatment for any reason.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck, S.L., Spain
Locations (28):
- Spain (28):
  - Hospital Universitario Príncipe de Asturias, Alcalá de Henares, Madrid
  - Hospital General de Alicante, Alicante
  - Hospital Nostra Senyora de Meritxell, Andorra
  - Hospital San Agustin, Avilés
  - Hospital San Agustín, Avilés
  - Hospital Materno Infantil de Badajoz, Badajoz
  - Hospital de Cruces-Baracaldo, Barakaldo
  - Hospital Sagrado Corazón, Barcelona
  - Hospital Puerta del Mar de Cádiz, Cadiz
  - Hospital Comarcal de Don Benito, Don Benito
  - Hospital de Elche, Elche
  - Hospital General de Elda, Elda
  - Hospital Clínico San Cecilio, Granada
  - Hospital SAS Jerez de la Frontera, Jerez de la Frontera
  - Hospital Severo Ochoa, Leganés, Madrid
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Hospital Univ. La Paz, Madrid
  - Hospital Materno Infantil de, Málaga
  - Hospital Virgen de la Arrixaca, Murcia
  - Hospital Central de Asturias, Oviedo
  - Hospital Son Espases, Palma de Mallorca
  - Hospital Virgen del Camino, Pamplona
  - Hospital Sant Joan de Reus, Reus
  - Hospital Parc Taulí de Sabadell, Sabadell
  - Hospital Clínico de Salamanca, Salamanca
  - Hospital Clínico Universitario, Santiago
  - Hospital de Valme. Seville, Seville
  - Hospital Virgen Macarena, Seville